CLINICAL TRIAL: NCT07359183
Title: Long Term Outcomes Associated With Attainment of Remission Following Oral Immunotherapy to Peanut, Egg and Cow's Milk (LPEM Study)
Brief Title: A Long Term, Observational Follow-Up Study of Children and Young People Who Underwent an 18-Month Course of Oral Immunotherapy Treatment for Peanut, Egg or Milk Allergy (5-15 Years Post-Treatment)
Acronym: LPEM
Status: Recruiting | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 121398
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Food Allergies; Peanut Allergies; Egg Allergy; Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Egg Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood - plasma and peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the long-term outcomes of children and young people who underwent an 18-month course of oral immunotherapy (OIT) treatment for peanut, egg or milk allergy. It aims to:

• Compare long-term changes in health-related quality of life (HRQL) at 5-15 years after stopping OIT in participants who achieved remission and those who did not.

Participants will attend a single follow-up visit for:

* A blood test
* Skin prick test (SPT)
* Allergy questionnaires

DETAILED DESCRIPTION:
The study population will be made up of participants from four clinical trials: PEAT, PrEMO, PPOIT-001 and PPOIT-002. They are being invited to participate in the LPEM observational study to evaluate the long-term outcomes of OIT.

* PEAT: Egg OIT. These participants are from the PEAT parent study (double-blind placebo-controlled randomized trial of probiotic and egg OIT).
* PrEMO: Egg or Milk OIT. These participants are from the PrEMO parent study (open label study of probiotic and egg and cow's milk OIT).
* PPOIT-001: Peanut OIT. These participants are from the PPOIT-001 parent study (double-blind placebo-controlled randomized trial of probiotic and peanut OIT).
* PPOIT-002: Peanut OIT. These participants are from the PPOIT-002 parent study (open label study of probiotic and peanut OIT).

Participants will have a blood sample taken at the visit to measure their peanut/egg/milk specific immunoglobulin E (sIgE) level. Plasma and peripheral blood mononuclear cells (PBMC) will also be stored for future analysis. A maximum of 50 milliliters (mL) of blood will be collected via venipuncture. If collection of blood via venipuncture is not possible, capillary blood via fingerprick technique will be collected instead (in which case only blood for the sIgE level will be collected, due to volume).

Participants will have a skin prick test completed at the visit to measure their allergy status. The skin prick test will include the following extracts:

* Positive control (histamine)
* Negative control (saline)
* House Dust Mite
* Rye Grass
* Peanut, Egg or Milk (depending on the participant's OIT treatment received in the parent study)

ELIGIBILITY:
Inclusion Criteria:

* Previous participant of PEAT, PrEMO, PPOIT-001 or PPOIT-002 parent study
* Received at least one dose of OIT treatment in the parent study
* Written informed consent from participant and/or parent/guardian (if below 18 years of age)

Exclusion Criteria:

-Have any conditions that, in the opinion of the investigator, precludes participation for reason of safety

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 147 participants will be recruited from the PEAT, PrEMO, PPOIT-001 and PPOIT-002 studies (Melbourne participants only), who received at least one dose of OIT.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Changes in health-related quality of life (HRQL) scores from baseline to 5-15 years after stopping oral immunotherapy (OIT) in individuals who achieved remission and those who did not, as measured by Food Allergy Quality of Life Questionnaires (FAQLQ). | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  HRQL scores were collected via validated surveys (FAQLQ) during the parent studies (PEAT, PrEMO, PPOIT-001 and PPOIT-002), and will be used again in this study for comparison. Changes in HRQL scores from the parent study (baseline) to 5-15 years after stopping OIT will be compared between the clinical outcome groups (Allergic or Sustained Unresponsiveness (SU)/Remission), as determined by the clinical outcome achieved at the end of treatment in the parent study. HRQL scores (reported as mean and standard deviation) will compare changes between the clinical outcome groups using generalised linear modules, adjusted for continuous variables as well as baseline HRQL scores. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test.

SECONDARY OUTCOMES:
Changes in HRQL scores from baseline to 5-15 years after stopping OIT in individuals who received OIT and those who received OIT placebo, as measured by FAQLQ. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  HRQL scores were collected via validated surveys (FAQLQ) during the parent studies (PEAT, PrEMO, PPOIT-001 and PPOIT-002), and will be used again in this study for comparison. Changes in HRQL scores from the parent study (baseline) to 5-15 years after stopping OIT will be compared between the treatment groups (OIT or placebo), as determined by the treatment group allocated in the parent study. HRQL scores (reported as mean and standard deviation) will compare changes between the treatment groups using linear regression adjusted for baseline HRQL scores. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test.
The incidence and severity of allergic reactions (in the preceding 12 months) at 5-15 years after stopping OIT in individuals who achieved remission and those who did not, as measured by REDCap Allergen Specific Questionnaire. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  Participants will complete a REDCap Allergen Specific Questionnaire indicating the number (0, 1, 2, 3, 4, 5, more than 5) of allergic reactions they experienced in the preceding 12 months to the allergen they received OIT treatment for in the parent study (peanut, egg or milk). In this REDCap Allergen Specific Questionnaire, participants will also indicate the number of times an Adrenaline Autoinjector was required for the management of the allergic reaction/s (0, 1, 2, 3, 4, 5, more than 5) in the preceding 12 months. Comparisons (reported as mean and standard deviation) will be made between the clinical outcome groups (Allergic or Sustained Unresponsiveness (SU)/Remission), as determined by the clinical outcome achieved at the end of treatment in the parent study. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test
The incidence and severity of allergic reactions (in the preceding 12 months) at 5-15 years after stopping OIT in individuals who received OIT and those who received OIT placebo, as measured by REDCap Allergen Specific Questionnaire. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  Participants will complete a REDCap Allergen Specific Questionnaire indicating the number (0, 1, 2, 3, 4, 5, more than 5) of allergic reactions they experienced in the preceding 12 months to the allergen they received OIT treatment for in the parent study (peanut, egg or milk). In this REDCap Allergen Specific Questionnaire, participants will also indicate the number of times an Adrenaline Autoinjector was required for the management of the allergic reaction/s (0, 1, 2, 3, 4, 5, more than 5) in the preceding 12 months. Comparisons (reported as mean and standard deviation) will be made between the treatment groups (OIT or placebo), as determined by the treatment group allocated in the parent study. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test.
Patterns of food ingestion (in the preceding 12 months) at 5-15 years after stopping OIT in individuals who achieved remission and those who did not, as measured by REDCap Allergen Specific Questionnaire. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  Participants will complete a REDCap Allergen Specific Questionnaire indicating ingestion in the preceding 12 months (yes/no) of the allergen they received OIT treatment for in the parent study (peanut, egg or milk). Comparisons (reported as absolute and relative frequencies) will be made between the clinical outcome groups (Allergic or Sustained Unresponsiveness (SU)/Remission), as determined by the clinical outcome achieved at the end of treatment in the parent study. Categorical outcomes such as allergen intake (yes/no) will be summarised as the number and proportion of subjects by clinical outcome group.
Changes in immunological markers from baseline to 5-15 years after stopping OIT in individuals who achieved remission and those who did not, as measured by allergen specific immunoglobulin E (sIgE) blood levels. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  Allergen specific immunoglobulin E (sIgE) blood levels were collected during the parent studies (PEAT, PrEMO, PPOIT-001 and PPOIT-002) and will be collected again in this study for comparison. Changes (reported as mean and standard deviation) in sIgE blood levels from the parent study (baseline) to 5-15 years after stopping OIT will be compared between the clinical outcome groups (Allergic or Sustained Unresponsiveness (SU)/Remission), as determined by the clinical outcome achieved at the end of treatment in the parent study. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test.
Changes in immunological markers from baseline to 5-15 years after stopping OIT in individuals who received OIT and those who received OIT placebo, as measured by allergen specific immunoglobulin E (sIgE) blood levels. | A single study visit (approximately 2 hours) will be conducted at 5-15 years after the participant completed OIT in their parent study.
  Allergen specific immunoglobulin E (sIgE) blood levels were collected during the parent studies (PEAT, PrEMO, PPOIT-001 and PPOIT-002) and will be collected again in this study for comparison. Changes (reported as mean and standard deviation) in sIgE blood levels from the parent study (baseline) to 5-15 years after stopping OIT will be compared between the treatment groups (OIT or placebo), as determined by the treatment group allocated in the parent study. If continuous outcomes do not follow normal distribution they will be summarised as median and interquartile ranges (IQR), and comparison between the groups will be performed using the Wilcoxon rank-sum (Mann-Whitney) test.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Chebar Lozinsky Rolnik, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected and stored in such a way that they can be used in future research projects. After 24 months following analysis and article publication, data may be made available for long-term use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access (including any conditions relating to MCRI's intellectual property).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months following analysis and article publication
Access Criteria: Data will be collected and stored in such a way that they can be used in future research projects. After 24 months following analysis and article publication, data may be made available for long-term use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access (including any conditions relating to MCRI's intellectual property).
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre